CLINICAL TRIAL: NCT03301818
Title: Vaginal Elasticity Assessment Before and After the Affect of Surgical Repair for Urinary Stress Incontinence (USI) on Vaginal Elasticity as Measured by Vaginal Tactile Imaging.
Brief Title: Vaginal Elasticity Assessment Before and After Surgical Repair for Urinary Stress Incontinence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0300-17-RMB
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing USI repair (Experimental)
  Interventions: Device: Vaginal tactile imager

INTERVENTIONS:
Device: Vaginal tactile imager — Patients will undergo elasticity assessment with vaginal tactile imaging the be once before surgical repair and twice after during a 3 month interval.

SUMMARY:
Female patients with USI will be evaluated for vaginal elasticity using vaginal tactile imaging both before and after surgery for the repair of the USI. Surgical repair will be performed by a single surgeon who will perform a tension free vaginal tape obturator (TVT-O) repair.

DETAILED DESCRIPTION:
Patients will be recruited and sign a consent form. The patients included are patients with USI that are candidates for a TVT-O repair.

Assessment of vaginal elasticity via vaginal tactile imaging will be performed at 3 different points:

* The day of surgery before surgery.
* The day after surgery.
* 3 months post-operational. Every patient will serve as her own control. Demographic, gynecologic and obstetric history will be obtained from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Any woman undergoing USI repair.

Exclusion Criteria:

* Women with high grade pelvic floor prolapse.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female.
Enrollment: 23 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Vaginal elasticity assessment | up to 3 months from enrollment
  Vaginal elasticity as measured by the vaginal tactile imager

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No